CLINICAL TRIAL: NCT01332851
Title: Training Social Work Providers: Intervention for Maltreating Families of Infants
Brief Title: Supporting Parents Program: Intervention for Families in CPS
Acronym: SPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Monica Oxford, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-103010-S; 1R01HD061362-01A2 (NIH)
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Child Abuse; Child Neglect
Keywords: child welfare; child protective services; child abuse; child neglect; infant; parenting
MeSH Terms: interventions — Health Resources; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Promoting First Relationships (PFR) (Experimental): PFR is a strengths-based 10 week in-home parenting intervention based on attachment theory. Each week has a theme for discussion, an activity, and time for "joining" - checking in with the parent, listening to their concerns and establishing a positive, supportive relationship. The sessions include handouts which focus on the content area covered that day and applying a topic to their relationship with their child. The provider also videotapes playtime between parent and child. On alternate weeks, the provider watches the video with the parent, reflecting on both the parent's and the child's needs. The provider helps the parent develop greater empathy and understanding of the child's needs and feelings, and helps the parent identify her own feelings and needs around parenting.
  Interventions: Behavioral: Promoting First Relationships (PFR)
- Resource & Referral (Active Comparator): This condition consists of 1) Resource and Referral assistance provided over the phone, and 2) Local Services Resource Packet. The participant receives a phone call from a Resource and Referral Specialist to conduct a needs assessment to identify the particular needs or concerns of the family (such as housing needs, mental health, tangible goods). If a need is identified, the Referral and Referral Specialist will provide the family with local information regarding the stated need. The R&R provider makes two follow-up check in calls with the families. In addition, families can call the Research and Referral Specialist if additional needs arise. The resource packet includes information organized by type of need or resource. These packets are updated regularly as services change over time.
  Interventions: Behavioral: Resource and Referral

INTERVENTIONS:
Behavioral: Promoting First Relationships (PFR) — PFR is a parenting intervention based on attachment theory and is strengths based. It is a 10 week intervention that is delivered in the home of the family.
  Arms: Promoting First Relationships (PFR)
Behavioral: Resource and Referral — Needs assessment, followed with a resource packet sent by mail
  Arms: Resource & Referral

SUMMARY:
The study evaluates the feasibility and effectiveness of a well-documented relationship-based intervention (Promoting First Relationships), compared to a resource and referral condition, in improving outcomes for families of infants and toddlers referred to Child Protective Services (CPS) for maltreatment. In addition, it evaluates the effectiveness of training community social service workers in providing the intervention.

DETAILED DESCRIPTION:
Child maltreatment has well-established, wide-ranging, and long-term negative effects on children. Most children who have experienced maltreatment and are receiving services through the Child Welfare System (CWS) remain in their homes with their caregivers. While the need for parenting services is extensive, few intervention programs have proven to be efficacious in reducing child abuse and neglect within the CWS population, especially for infants and toddlers. It is essential that social service practitioners within the CWS delivery system are equipped to provide brief interventions to maltreating parents. This grant, "Training Social Work Providers: Intervention for Maltreating Families of Infants and Toddlers," is an evaluation of a training program for social welfare providers to implement a brief attachment theory-based intervention to families who have been investigated for child abuse and neglect by Child Protective Services. The program (Promoting First Relationships [PFR]; Kelly, Buehlman, & Caldwell, 2000) will be tested at two levels: through social welfare practice and at the level of outcomes for children and families.

Social service providers will be trained to deliver PFR to families under investigation for maltreatment by the Department of Social and Health Services, in two counties in Washington State. Subsequently, families under investigation by CPS will be recruited into the study and randomly assigned to the experimental group (receiving the PFR intervention) or to the comparison group (receiving resources and referrals).

The specific aims of this study are to (1) Test the effectiveness of training community social welfare service providers in the use of attachment-based interventions by measuring their pre-training and post-training service provision strategies and interactions with maltreating families; (2) To test the effects of a relationship and attachment-based intervention with infants/toddlers of parents identified as maltreating by comparing them to a control group on rates of re-referral to CPS, severity of referral, and foster care placement; and (3) To conduct a test of the effectiveness of an attachment-based intervention on child well-being by comparing experimental and comparison groups on important outcomes (attachment security, emotional regulation, behavior, and developmental functioning).

RELEVANCE Child maltreatment is a serious public health issue, affecting close to a million children nationally every year. The establishment of effective evidence-based interventions for high-risk families is essential to curtail the devastating long-term effects of maltreatment. The proposed study tests the feasibility and effectiveness of a well-documented relationship-based intervention (Promoting First Relationships) in improving outcomes for families referred to CPS for maltreatment.

ELIGIBILITY:
Inclusion Criteria:

* Biological parents and their child aged 10-24 months, who is an identified victim for referral to CPS, and who are parenting their child a majority of the time
* Families served by CPS offices in Snohomish and Skagit counties, in the state of Washington
* Families at moderate to high risk for maltreatment (physical abuse, neglect, or emotional maltreatment) and under investigation by Child Protective Services
* English speaking primary caregiver
* Telephone access
* Current housing

Exclusion Criteria:

* Experiencing an acute crisis (homelessness, hospitalization, imprisonment)
* Identified child (in a risk only CPS intake) or identified victim (in CPS intakes with allegations) has a voluntary services agreement within 2 weeks of a newly opened investigation
* Identified child (in a risk only CPS intake) or identified victim (in CPS intakes with allegations) has a dependency filing within 2 weeks of a newly opened investigation
* Previously received the Promoting First Relationships intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica L Oxford, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Family & Child Nursing, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oxford ML, Spieker SJ, Lohr MJ, Fleming CB. Promoting First Relationships(R): Randomized Trial of a 10-Week Home Visiting Program With Families Referred to Child Protective Services. Child Maltreat. 2016 Nov;21(4):267-277. doi: 10.1177/1077559516668274. Epub 2016 Sep 21. PMID 27646148
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219
- See also: Promoting First Relationships (PFR) — http://www.pfrprogram.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: DCFS volunteer scanned WA State DSHS database monthly (January 2011- January 2014); created list of possibly eligible families (N=1070). Potential participants contacted (n=556; n=514 unable to be contacted), permission received to forward their contact information to the study (n=251; n=172 ineligible, n=133 declined).
Pre-assignment Details: 4 participants were not randomized (2 already had the study intervention, 1 refused to sign the HIPAA agreement, and 1 was not located). 19 additional caregivers were enrolled post randomization when the study parent lost custody of their child. They were not "randomized" to a condition, but they were consented to participate and supplied data.
Groups:
- Promoting First Relationships (PFR): PFR is a parenting intervention based on attachment theory and is strengths based. It is a 10 week intervention that is delivered in the home. Each week has a theme for discussion, an activity which includes videotaping or viewing and reflecting on a videotaped session, and time for "joining" - checking in with the parent, listening to their concerns and establishing a positive, supportive relationship. The sessions include handouts which focus on the content area covered that day and applying a topic to their relationship with their child. The provider also videotapes playtime between parent and child. On alternate weeks, the provider watches the video with the parent, reflecting on both the parent's and the child's needs. The provider helps the parent develop greater empathy and understanding of the child's needs and feelings, and helps the parent identify her own feelings and needs around parenting.
- Resource & Referral (R&R): This condition consists of 1) Resource and Referral personal assistance provided over the phone, and 2) Local Services Resource Packet. The participant receives a phone call from a Resource and Referral Specialist hired by the project. The service consists of a needs assessment to identify the particular needs or concerns of the family (such as housing needs, mental health, tangible goods). If a need is identified, the Referral and Referral Specialist will provide the family with local information regarding the stated need (such as a phone number to a housing assistance program, location of local food bank). The R&R provider makes two follow-up check in calls with the families. In addition, families can call the Research and Referral Specialist if additional needs arise. The resource packet includes information organized by type of need or resource. These packets are updated regularly as services change over time.
Period: Overall Study
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Started | 124 | 123
Completed Intervention (Intent-to-treat: we attempted to retain all participants, regardless of intervention completion.) | 107 (9 no intervention, 8 <full dose, 107 full dose; 3 new caregivers enrolled-initial parent dropped out) | 110 (4 no intervention, 9 <full dose, 110 full dose; 4 new caregivers enrolled-initial parent dropped out)
Completed Follow up 1 (Attempted to retain all participants regardless of intervention completion) | 116 | 112 (Includes 1 new caregiver enrolled due to initial parent no longer parenting)
Completed Follow up 2 (Attempted to retain all participants regardless of intervention and/or follow up 1 completion) | 111 (Includes 1 new caregiver enrolled due to initial parent no longer parenting) | 111 (Includes 4 new caregivers enrolled due to initial parent no longer parenting)
Completed Follow up 3 (Attempted to retain all participants regardless of intervention and/or follow up 1 & 2 completion) | 113 (Includes 3 new caregivers enrolled due to initial parent no longer parenting) | 110 (Includes 3 new caregivers enrolled due to initial parent no longer parenting)
Completed | 113 | 110
Not Completed | 11 | 13
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Promoting First Relationships (PFR): PFR is based on attachment theory and is strengths based. The 10 week intervention is delivered in the home of the family. Each week has a theme for discussion, an activity which includes videotaping or viewing and reflecting on a videotaped session, and time for "joining" - checking in with the parent, listening to their concerns and establishing a positive, supportive relationship. The sessions include handouts, one with the content area covered that day and one applying a topic to their relationship with their child. The provider also videotapes playtime between parent and child and alternates every other week with watching the video with the parent. When the parent and provider watch the video of the previous session, they reflect about what the needs are of both the parent and the child. The provider helps the parent develop greater empathy and understanding of the child's needs and feelings, and helps the parent identify her own feelings and needs around parenting.
- Resource & Referral: This condition will consist of 1) Resource and Referral Personal Assistance provided over the phone, and 2) Local Services Resource Packet. The participant in this arm of the intervention trial receive a phone call from a Resource and Referral Specialist hired by the project. The service consists of a needs assessment to identify the particular needs or concerns of the family (such as housing needs, mental health, tangible goods). If a need is identified, the Referral and Referral Specialist will provide the family with local information regarding the stated need (such as a phone number to a housing assistance program, location of local food bank). In addition, families in this condition will have the Research and Referral Specialist's phone number they can call if an additional need arises. The resource packet will include information organized by type of need or resource. These packets will be updated regularly as services change over time.
- Total: Total of all reporting groups
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral | Total
Number analyzed (Participants) | 124 | 123 | 247
Age, Continuous [Mean (Standard Deviation); unit: years]
  parent age in years | 26.41 (5.19) | 27.04 (6.25) | 26.72 (5.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Parent gender: Female | 112 | 113 | 225
  Parent gender: Male | 12 | 10 | 22
Region of Enrollment [Number; unit: participants] — All 247 parents were recruited from Snohomish, southern Skagit, and northern King Counties, Washington, USA
  participants
    United States | 124 | 123 | 247

OUTCOME MEASURES:

1. Primary Outcome: Child Welfare Outcomes: CWS Removal From Birth Parent Home
Description: Official child welfare administrative records indicating whether child was removed from the birth parent home within one year of parent completing intervention (or one year after estimated date intervention would have been completed, for parents who did not complete). Data were analyzed with a survival model that predicted hazard of being removed from the birth parent home.
Time Frame: 1 year post intervention
Measure: Number; unit: participants
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral
Number analyzed (Participants) | 124 | 123
participants | 7 | 16
Statistical Analysis 1: Comparison: Promoting First Relationships (PFR) vs Resource & Referral; Child welfare system removals were analyzed with a survival models that used condition assignment to predict hazard of being removed from the birth parent home; Test type: Superiority; p = .043, Regression, Cox — We used a threshold of p < .05 as the criterion for statistical significance; Cox Proportional Hazard = 2.50, 95% CI 2-sided [1.03 to 6.10] — The hazard ratio of 2.5 indicates that children with parents in the control group were 2.5 times more likely to be removed from their home and placed into foster care compared to the intervention group

2. Primary Outcome: Parental Sensitivity (Video Recorded Observation Coded by Blind Coders)
Description: Parent sensitivity was measured at all four time points by a modified total score of the Nursing Child Assessment Teaching Scale (NCATS; Barnard, 1994), a videotaped interaction to assess caregiver sensitivity, stimulation of the child, and emotional responsiveness during interaction were scored. The scale was modified to exclude some items from the original measure that demonstrated low variability in other studies. A total score was based on 45 items, possible range 0 - 45. Items covered mutuality (e.g. contingency, gaze, and positive affect), caregiver verbal and nonverbal support of child, and sensitive instruction during the teaching task. Items were scored yes (1) or no (0), and yes scores were summed. Cronbach's alpha for the sensitivity scale ranged from .68 to .72. A single, blinded coder was trained to reliability by a certified NCATS instructor and passed regular reliability checks. Higher scores indicate greater parental sensitivity.
Time Frame: Baseline, post intervention (approximately 4 months from baseline, 3 month follow up (~7 months from baseline), 6 month follow up (~ 10 months from baseline)
Population: ITT, all 247 parents were coded on the sensitivity measure and were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Promoting First Relationships (PFR): Assigned to Promoting First Relationships (PFR) condition
- Resource & Referral: Assigned to Resource and Referral condition
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral
Number analyzed (Participants) | 124 | 123
units on a scale
  Baseline | 26.94 (4.22) | 27.97 (4.71)
  post intervention | 27.34 (4.97) | 26.70 (4.63)
  3 month fu | 27.77 (4.54) | 27.39 (4.59)
  6 month fu | 28.07 (4.31) | 27.18 (5.20)
Statistical Analysis 1: Comparison: Promoting First Relationships (PFR) vs Resource & Referral; Mixed models were estimated in which post-intervention scores were nested. The intercept (representing the average score across post-intervention time points) was modeled as having a random effect. The intercept in the mixed model was regressed on intervention condition (R&R = 0, PFR = 1), baseline sensitivity score, months between baseline and end of intervention, and age of child at baseline; Test type: Superiority or Other; p < .05, Mixed Models Analysis; Mean Difference (Net) = 0.94, Standard Error of Mean 0.42 — Parents in the PFR condition were 0.94 higher on sensitivity scores (on the unstandardized sensitivity measure) across the three post-intervention time points than parents in the R&R condition. The standard error (SE) of this difference was .42

3. Primary Outcome: Secure Base Behavior (Observation During Research Visit; Higher Score Indicates Greater Security)
Description: Secure base behavior was measured with the Toddler Attachment Sort-45 (TAS-45; Kirkland, Bimler, Drawneek, McKim, & Schölmerich, 2004). The TAS-45 is based on 39 items from the Attachment Q-Sort (AQS; Waters, 1987), an attachment measure that has been extensively validated (van IJzendoorn, Vereijken, Bakermans-Kranenburg, & Riksen-Walraven, 2004), plus six items tapping atypical affective communication. After home visits, research visitors sorted cards for 45 descriptive statements of child attachment behavior into five piles representing "most like" to "least like" the child. Item scores were standardized within individuals and then compared to a security profile to arrive at an security score. Higher value indicates greater secure base behavior. Because scores are based standardized item scores weighted by proximity to the secure profile, the possible range is large, difficult to determine, and not reported in the instrument manual. The observed range was from -.62 to +1.00.
Time Frame: as for outcome 2
Population: All 247 children in the study were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral
Number analyzed (Participants) | 124 | 123
units on a scale
  Baseline | .45 (.36) | .46 (.34)
  Post Intervention | .52 (.35) | .51 (.35)
  3 month follow up | .56 (.32) | .56 (.34)
  6 month follow up | .62 (.33) | .57 (.31)
Statistical Analysis 1: Comparison: Promoting First Relationships (PFR) vs Resource & Referral; Mixed models were estimated in which post-intervention scores were nested. The intercept (representing the average score across post-intervention time points) was modeled as having a random effect. The intercept in the mixed model was regressed on intervention condition (R&R = 0, PFR = 1), baseline security score, months between baseline and end of intervention, and age of child at baseline; Test type: Superiority; p > .05, Mixed Models Analysis; Mean Difference (Net) = .05, Standard Error of Mean .03 — The PFR group had a higher mean compared to the R&R group. (the absolute value of the standardized effect is d=.15)

4. Secondary Outcome: Parenting Stress: Dysfunctional Interaction
Description: Parenting stress was measured by scales selected from the Parenting Stress Index and the Parenting Stress Index-Short Form (PSI-3, PSI-SF; Abidin, 1995). The Parent-Child Dysfunctional Interaction Scale from the PSI-SF (11 items). Items were rated on 4-point scales (strongly agree to strongly disagree). Two items measuring parental educational attainment from the original parenting competence scale were omitted due to excessive missing data. Higher scores indicate greater parental stress associated with feelings of dysfunctional parent-child interactions (i.e., interactions are not reinforcing or satisfying). Alphas ranged from .71-.94 across time points. Possible range 11-55, observed range 12 to 43.
Time Frame: Baseline, post intervention (approximately 4 months from baseline, 3 month follow up from post intervention (~7 months from baseline), 6 month follow up (~ 10 months from baseline)
Population: ITT: All 247 parents were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 124 | 123
units on a scale
  Baseline | 18.44 (5.28) | 18.60 (5.67)
  3-month post-intervention follow-up | 18.48 (5.73) | 18.80 (5.04)
  6-month post-intervention follow-up | 21.26 (4.78) | 21.70 (5.26)
Statistical Analysis 1: Comparison: Promoting First Relationships (PFR) vs Resource & Referral (R&R); Mixed models were estimated in which post-intervention scores were nested. The intercept (representing the average score across post-intervention time points) was modeled as having a random effect. The intercept in the mixed model was regressed on intervention condition (R&R = 0, PFR = 1), baseline problem behavior score, months between baseline and end of intervention, and age of child at baseline; Test type: Superiority; p > .05, Mixed Models Analysis; Mean Difference (Net) = -.20, Standard Error of Mean .50 — The adjusted mean across the two post-intervention time points was -.20 (SE=.50) lower in the PFR group than R&R group. The standardized effect size was d=.04

5. Secondary Outcome: Parent Stress: Competence (Higher Score Means More Stress)
Description: At baseline, 3-month post-intervention follow-up, and 6-month post-intervention follow-up, parenting stress was measured by scales selected from the Parenting Stress Index and the Parenting Stress Index-Short Form (PSI-3, PSI-SF; Abidin, 1995). The Parenting Competence Scale from the PSI-3 (11 items) was used. Items were rated on 4-point scales (strongly agree to strongly disagree). Two items measuring parental educational attainment from the original parenting competence scale were omitted due to excessive missing data. Higher scores indicate greater parental stress associated with feelings of incompetence. Alphas ranged from .71-.94 across time points. Possible range 11 - 55, observed range 11 - 39.
Time Frame: Baseline 3-month post-intervention (~7 months post baseline), 6-month follow up (~ ten months post baseline)
Population: ITT: All 247 parents were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 124 | 123
units on a scale
  Baseline | 16.03 (4.75) | 16.59 (5.21)
  3-month post-intervention follow-up | 19.73 (6.52) | 19.95 (6.07)
  6-month post-intervention follow-up | 19.80 (6.54) | 19.33 (6.03)
Statistical Analysis 1: Comparison: Promoting First Relationships (PFR) vs Resource & Referral (R&R); Mixed models were estimated in which post-intervention scores were nested. The intercept (representing the average score across post-intervention time points) was modeled as having a random effect. The intercept in the mixed model was regressed on intervention condition (R&R = 0, PFR = 1), baseline competence stress score, months between baseline and end of intervention, and age of child at baseline; Test type: Superiority; p > .05, Mixed Models Analysis; Mean Difference (Net) = .41, Standard Error of Mean .53 — The adjusted mean across post-intervention time points was .41 (SE=.53) higher in the PFR group than the R&R group. The standardized effect size was d=-.07

6. Secondary Outcome: Child Social Emotional Development (Higher Scores Indicate More Competence)
Description: Child social-emotional competence (11 items; alphas = .69-.70) was measured by the Brief Infant Toddler Social and Emotional Assessment (BITSEA; Briggs-Gowan & Carter, 2002). Possible range is 0 - 22. Parent report of child social-emotional competence in the last month were rated on a 3-point scale (not true/rarely; somewhat true/sometimes; very true/often). Higher scores indicate more competence.
Time Frame: as for outcome 2
Population: ITT: All 247 children were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 124 | 123
units on a scale
  Baseline | 15.80 (3.30) | 16.30 (3.56)
  Post-intervention | 17.40 (3.10) | 17.37 (2.93)
  3-month follow-up | 17.55 (2.90) | 17.41 (2.93)
  6-month follow-up | 17.72 (2.81) | 17.78 (2.95)
Statistical Analysis 1: Comparison: Promoting First Relationships (PFR) vs Resource & Referral (R&R); Mixed models were estimated in which post-intervention scores were nested. The intercept (representing the average score across post-intervention time points) was modeled as having a random effect. The intercept in the mixed model was regressed on intervention condition (R&R = 0, PFR = 1), baseline social-emotional competence score, months between baseline and end of intervention, and age of child at baseline; Test type: Superiority; p > .05, Mixed Models Analysis; Mean Difference (Net) = .24, Standard Error of Mean .25 — The PFR group had a higher mean level of social and emotional development compared to the R&R group (the absolute value of the standardized effect is d=.10)

7. Secondary Outcome: Child Behavior Problems
Description: Child behavior problems (31 items; alphas =.77-.79) were measured by parent report on the Brief Infant Toddler Social and Emotional Assessment (BITSEA; Briggs-Gowan & Carter, 2002). Descriptions of positive and problematic social-emotional behaviors in the last month were rated on a 3-point scale (not true/rarely; somewhat true/sometimes; very true/often; items score 0, 1, 2 respectively). Higher score indicates more child behavior problems as noted by the parent. Possible range is 0 - 62.
Time Frame: as for outcome 2
Population: ITT: all 247 children were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 124 | 123
units on a scale
  Baseline | 10.84 (5.79) | 10.96 (6.47)
  Post-intervention | 11.01 (6.12) | 12.19 (7.08)
  3-month follow-up | 11.82 (6.60) | 11.80 (7.75)
  6-month follow-up | 11.23 (7.51) | 11.87 (8.43)
Statistical Analysis 1: Comparison: Promoting First Relationships (PFR) vs Resource & Referral (R&R); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p > .05, Mixed Models Analysis; Mean Difference (Net) = -.80, Standard Error of Mean .66 — The PFR group had lower mean level of problem behavior compared to the R&R group (the absolute value of standardized effect is d= .12)

8. Secondary Outcome: Child Emotion Regulation
Description: Bayley Behavior Ratings (Bayley, 1993) to assess emotion regulation. At baseline and again at the 3-month follow-up, blinded research visitors rated the child's behavior during administration of a standardized developmental test using the Bayley Behavior Rating Scales (BRS; Bayley 1993). Seven items in the BRS comprise the emotion regulation scale and capture how well the child adapts to challenging stimuli and frustration (alphas = .79-.83). Possible range is 1 - 5, the mean of seven items scored from 1 to 5. Higher scores indicate better emotional regulation.
Time Frame: Baseline and at the 3 month follow up (~ 7 months post baseline)
Population: ITT: all 247 children were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 124 | 123
units on a scale
  Baseline | 3.73 (.66) | 3.80 (0.60)
  3-month post-intervention follow-up | 3.82 (.64) | 3.96 (0.65)
Statistical Analysis 1: Comparison: Promoting First Relationships (PFR) vs Resource & Referral (R&R); Tested mean differences by condition at 3-month follow-up controlling for baseline score, months between baseline and the end of the intervention, and age of child and using an ANVOVA/regression model. Null hypothesis was that post-intervention means were equal; Test type: Superiority; p > .05, Regression, Linear; Mean Difference (Net) = -.07, Standard Error of Mean .08 — Adjusted mean at 3-month post-intervention was -.07 (SE=.08) lower for PFR compared to R&R group

9. Secondary Outcome: Child Engagement/Exploration
Description: At baseline and again at the 3-month follow-up, blinded research visitors rated the child's behavior during administration of a standardized developmental test using the Bayley Behavior Rating Scales (BRS; Bayley 1993). Engagement/exploration consists of six items rated for exploratory behavior in the testing situation (alphas = .75-.76). The items were scored on a rage of 1 to 5, the mean of the six items was computed and the possible range is 1 to 5. Higher scores indicate more engagement.
Time Frame: Baseline and at the 3 month follow up (~ 7 months post baseline)
Population: ITT: all 247 children were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 124 | 123
units on a scale
  Baseline | 4.19 (.63) | 4.21 (.55)
  3-month post-intervention follow-up | 4.15 (.57) | 4.25 (.58)
Statistical Analysis 1: Comparison: Promoting First Relationships (PFR) vs Resource & Referral (R&R); Test type: Superiority; p > .05, Regression, Linear; Mean Difference (Net) = -.06, Standard Error of Mean .08 — Adjusted mean at 3-month post-intervention was -.06 (SE=.08) lower for PFR compared to R&R group

10. Secondary Outcome: Child Atypical Affective Communication (Observation)
Description: Atypical, affective communication were measured with the Toddler Attachment Sort-45 (TAS-45; Kirkland, Bimler, Drawneek, McKim, & Schölmerich, 2004). The TAS-45 is based on 39 items from the Attachment Q-Sort (AQS; Waters, 1987), an attachment measure that has been extensively validated (van IJzendoorn, Vereijken, Bakermans-Kranenburg, & Riksen-Walraven, 2004), plus six additional items tapping atypical, affective communication. Immediately after research home visits, the research visitors sorted cards for 45 descriptive statements of child attachment behavior into five piles representing "most like" to "least like" the child. Item scores were standardized within individuals and then scaled with weights for the D hotspot. Because scores are based on standardized item scores, the possible range is large, difficult to determine, and not reported in the instrument manual. Observed range -1.511 to + .860.
Time Frame: as for outcome 2
Population: ITT: all 247 children were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 124 | 123
units on a scale
  Baseline | -.91 (.47) | -.94 (.44)
  Post-intervention | -.96 (.42) | -.92 (.42)
  3-month follow-up | -1.02 (.36) | -1.00 (.38)
  6-month follow-up | -1.05 (.33) | -.99 (.34)
Statistical Analysis 1: Comparison: Promoting First Relationships (PFR) vs Resource & Referral (R&R); Mixed models were estimated in which post-intervention scores were nested. The intercept (representing the average score across post-intervention time points) was modeled as having a random effect. The intercept in the mixed model was regressed on intervention condition (R&R = 0, PFR = 1), baseline score, months between baseline and end of intervention, and age of child at baseline; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Net) = -.07, Standard Error of Mean .04 — The PFR group had lower atypical affective communication compared to the R&R group (the absolute value of the standardized effect size was d=.19)

11. Secondary Outcome: Parent-Child Interaction (Video Recorded Observation Coded by Blind Coders)
Description: Coding Interactive Behavior-Child & Parent Outcomes (CIB; Feldman, 1998). Parent-child 10-minute free play interaction coded for child social engagement, child negative affect, and dyadic reciprocity; parental sensitivity and reciprocity, parental intrusiveness, and parental withdrawal.
  NOTE: THIS MEASURE WAS COLLECTED AND CODED. HOWEVER, THE MEASURE SUFFERED FROM LOW INTERNAL CONSISTENCY AND RESTRICTED VARIATION (I.E., A LARGE PORTION OF SCORES WERE NEAR THE MAXIMUM POSSIBLE VALUE). WE DID COMPARE SCORES BY CONDITION AND ALL COMPARISONS INDICATED NONSIGNIFICANT DIFFERENCES BETWEEN PFR AND R&R CONDITIONS. DUE TO LOW RELIABILITY AND RESTRICTED VARIATION OF THE MEASURE, IT WAS DECIDED TO NOT REPORT THESE RESULTS.
Time Frame: as for outcome 2
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Parental Confidence
Description: Caregiving Helplessness Questionnaire (CHQ; George, Coulson, Majany, & Soloman, 1995) subscales: parent-child frightened and parent helplessness. NOTE: THIS MEASURE WAS COLLECTED AND COMPARISONS BETWEEN PFR AND R&R INDICATED NONSIGNIFICANT DIFFERENCES. DUE TO LOW INTERNAL CONSISTENCY OF THE MEASURE, IT WAS DECIDED TO NOT REPORT PFR VS. R&R COMPARISONS FOR THIS MEASURE.
Time Frame: as for outcome 2
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Parental Mindfulness
Description: "About My Baby": three open-ended questions; coded to assess "mindfulness" representations of the child's mental life. NOTE: THIS MEASURE WAS DROPPED FROM THE STUDY. OPEN-ENDED QUESTIONS WERE INCLUDED IN INITIAL ASSESSMENTS. ANSWERS WERE REVIEWED BY THE RESEARCH TEAM, AND IT WAS DECIDED THAT RELIABLE AND VALID CODING WAS NOT POSSIBLE.
Time Frame: as for outcome 2
Population: NOTE: THIS MEASURE WAS DROPPED FROM THE STUDY
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Maternal Unrealistic Expectations
Description: Parent Opinion Questionnaire (POQ; Azar et al., 1984): questionnaire to assess unrealistic parental expectations of child behavior in the areas of self-care, help and affection to parents, leaving children alone, proper feelings and behavior punishment, and family responsibility. NOTE: THIS MEASURE WAS COLLECTED. RESPONDENTS WERE OFFENDED BY SOME QUESTIONS, WE REDUCED THE NUMBER OF QUESTIONS AT BASELINE AND COLLECTED THE FULL INSTRUMENT AT FOLLOW UP 1. HOWEVER, IT SHOWED LIMITED VARIABILITY. COMPARISONS BETWEEN PFR AND R&R CONDITIONS INDICATED NONSIGNIFICANT DIFFERENCES. DUE TO THE LIMITED VARIABILITY, IT WAS DECIDED NOT TO REPORT THESE RESULTS.
Time Frame: Baseline and Post intervention (~ 4 months post baseline)
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral (R&R)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years post baseline
Arm/Group | Promoting First Relationships (PFR) | Resource & Referral
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/123
Other Adverse Events (participants affected / at risk) | 36/124 | 42/123
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Promoting First Relationships (PFR) (N=124) | Resource & Referral (N=123)
CPS reports (Investigations) | 36 (73) | 42 (69) — Allegation of maltreatment reported to Child Protective Services linked to the enrolled parent's target study child
Removal from home (Investigations) | 7 (7) | 16 (16) — Removal of the enrolled parent's target study child from birth parent home following CPS investigation

LIMITATIONS AND CAVEATS:
Generalizability limited by sample selection criteria. Follow-up was only 6-months post-intervention for most outcomes although child welfare records covered 1 year post-intervention. Parent report was used for some key outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No